CLINICAL TRIAL: NCT05128162
Title: A Phase 2a, Open-label, Pilot Study to Assess the Safety and Efficacy of Psilocybin Administration in Concert With Psychotherapy Among Adult Patients With Fibromyalgia
Brief Title: Open-label Study to Assess the Safety and Efficacy of Psilocybin With Psychotherapy in Adult Participants With Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kevin Boehnke (Other)
Responsible Party: Sponsor-Investigator, Kevin Boehnke, Research Assistant Professor, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00208367
Record Dates: First submitted 2021-10-14; First posted 2021-11-19 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Psilocybin; Psychotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label Oral Psilocybin (Experimental): This is an open-label study, and participants who meet the inclusion and exclusion criteria will be eligible and invited to enroll. Enrolled participants are planned to receive 2 doses of psilocybin: a 15 mg dose followed 2 weeks later by a 25 mg dose. The total planned duration of the study for an individual participant from screening to last follow-up is approximately 8 months.
  Interventions: Drug: Psilocybin; Behavioral: Psychotherapy

INTERVENTIONS:
Drug: Psilocybin — Two oral doses of psilocybin in a capsule formulation taken approximately 2 weeks apart.
Behavioral: Psychotherapy — 1. Pre-dose preparatory sessions; 2. Dosing day monitoring; and, 3. Post-dose integration sessions.

SUMMARY:
The pressing need for effective fibromyalgia (FM) treatments, the known safety of psilocybin therapy, and the mechanistic plausibility for potential benefit provide a backdrop for investigating psilocybin therapy as a treatment for FM. The primary objective of this study is to evaluate the clinical benefit of oral psilocybin in concert with psychotherapy to treat chronic pain symptoms in patients with FM.

DETAILED DESCRIPTION:
Fibromyalgia is a chronic syndrome of widespread musculoskeletal pain that often manifests with a cluster of co-occurring symptoms, including sleep disturbances, fatigue, cognitive dysfunction, and mood problems including anxiety and depression. Recent studies have provided evidence of altered central pain pathways. Current management of FM typically takes a multidimensional approach including behavioral therapy, exercise, and medication. However, current medications provide only modest benefit and carry significant side effect burden, leading many people with FM to seek other alternatives.

Psilocybin therapy (psilocybin delivered in concert with psychotherapy) may be a potentially safe and effective treatment for symptoms associated with FM. Indeed, psilocybin therapy has shown positive effects in treating cancer-related psychiatric distress, depression and anxiety, treatment-resistant depression, and nicotine or alcohol addiction. The United States Food and Drug Administration (FDA) has granted a Breakthrough Therapy designation for psilocybin in treatment-resistant depression and major depressive disorder. Psilocybin therapy is generally safe and well-tolerated when conducted under controlled conditions. While no clinical studies have explored psychedelic effects among people with FM, a recent review outlined potential mechanisms through which psychedelics could alleviate chronic pain symptoms.

ELIGIBILITY:
Inclusion Criteria

Participants are eligible to be included in the study only if all of the following criteria apply:

Age

- Participant must be 25 to 64 years of age, inclusive, at the time of signing the informed consent form.

Type of Participant and Disease Characteristics

* Participant must meet "criteria for FM per the 2016 FM survey criteria."
* Concurrent psychotherapy is allowed if the type and frequency of the therapy has been stable for at least 2 months prior to screening and is expected to remain stable during participation in the study.
* Participant must be a non-smoker (tobacco).
* Participant must be medically stable as determined by screening for medical problems via a personal interview and/or, a medical questionnaire, and an ECG, within 1 month of starting active intervention (performed during screening).
* Participant must agree to consume approximately the same amount of caffeine-containing beverage (e.g., coffee, tea, cola) that he/she consumes on a usual morning, before arriving at the research unit on the mornings of psilocybin session days. If the participant does not routinely consume caffeinated beverages, he/she must agree to not do so on psilocybin session days.
* Participant must agree to refrain from using any psychoactive drugs, including alcoholic beverages and nicotine, within 24 hours before and after each psilocybin administration. The exception is caffeine.
* Participant must agree to not take sildenafil (Viagra®), tadalafil, or similar medications within 72 hours before and after each psilocybin administration.
* Participant must agree to not take any pro re nata (PRN) medications on the mornings of psilocybin sessions.
* Participant must agree that for 7 days before each psilocybin session, he/she will refrain from taking any nonprescription medication, cannabis, nutritional supplement, or herbal supplement except when approved by the Principal Investigator. Exceptions will be evaluated by the Principal Investigator and will include acetaminophen, non-steroidal anti-inflammatory drugs, and common doses of vitamins and minerals.
* Participant must have at least a high school level of education or equivalent (e.g., General Educational Development [GED] Test).

Sex and Contraceptive/Barrier Requirements

* Contraceptive use by women and men should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

  1. Females of reproductive potential must agree to use effective birth control for the duration of active intervention (defined as the time from the Baseline [deep phenotyping] visit until the EOT [deep phenotyping] visit).
  2. Sexually active male participants and/or their female partners must agree to use effective birth control for the duration of active intervention (defined as the time from the Baseline [deep phenotyping] visit until the EOT [deep phenotyping] visit) of the male participant. Male participants must also agree not to donate sperm for the duration of active intervention.

     Informed Consent
* Participant has provided informed consent as described in Appendix 1, Section 10.1.3 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria

Participants are excluded from the study if any of the following criteria apply:

Medical Conditions

* Participant has had (within the past 1 year) a cardiovascular condition such as coronary artery disease, stroke, angina, uncontrolled hypertension, a clinically significant ECG abnormality (e.g., atrial fibrillation), prolonged QTc interval (i.e., QTc > 450 msec), artificial heart valve, or transient ischemic attack.
* Participant has epilepsy with a history of seizures.
* Participant has insulin-dependent diabetes.
* Participant is taking an oral hypoglycemic agent and has a history of hypoglycemia.
* Participant has active auto-immune disease (e.g., lupus, rheumatoid arthritis).
* Participant has a current or past history of meeting Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) criteria for schizophrenia spectrum or other psychotic disorders (except substance/medication-induced or due to another medical condition), or bipolar I or II disorder measured via SCID-5 and SCID-5-PD.
* Participant has a current or past history (within 1 year) of meeting DSM-5 criteria for a moderate or severe alcohol, tobacco, or other drug use disorder (excluding caffeine) measured via relevant questions from the SCID-5.
* Participant has a history of a medically significant suicide attempt.

Prior/Concomitant Therapy

* Participant is taking psychoactive prescription medication (e.g., opioids, tramadol, benzodiazepines) on a regular basis (i.e., more than 2 times a week).
* Participant is currently taking an antidepressant. Participants will also be required to refrain from using antidepressant medications through the completion of primary outcome assessments. Note: if a participant self-initiates a medication taper with the consent and support of their physician, they can re-screen after the appropriate time period.
* Participant is currently taking bupropion or antidepressants other than selective serotonin reuptake inhibitors (SSRIs), selective norepinephrine reuptake inhibitors (SNRIs).
* Participant is currently taking on a regular (e.g., daily) basis any medications having a primary centrally-acting serotonergic effect, including monoamine oxidase inhibitors (MAOIs). For individuals who have intermittent or PRN use of such medications, psilocybin sessions will not be conducted until at least 5 half-lives of the agent have elapsed after the last dose.
* Participant tests above 0.02% blood alcohol content on breath alcohol testing and/or positive for cocaine, methamphetamine, or opioids on urine drug testing.
* Participant has a psychiatric condition judged to be incompatible with establishment of rapport or safe exposure to psilocybin.

Prior/Concurrent Clinical Study Experience

- Participant is currently in another clinical trial.

Diagnostic assessments

* Participant has a significant suicide risk as defined by:

  1. suicidal ideation as endorsed on items 4 or 5 on the C-SSRS within the past year at Screening or at Baseline; or
  2. suicidal behaviors within the past year; or
  3. clinical assessment of significant suicidal risk during participant interviews
* Participant has severe depression as measured through PHQ-8 at Screening.

Other Exclusions

* Participant is pregnant (as indicated by a positive urine pregnancy test assessed at Screening and before each psilocybin session) or nursing.
* Participant is a WOCBP and sexually active, or a man and sexually active, and not practicing an effective means of birth control.
* Participant has a confirmed first- or second-degree relative with schizophrenia spectrum or other psychotic disorders (except substance/medication-induced or due to another medical condition), or bipolar I or II disorder.

Ages: 25 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin F Boehnke, PhD, Principal Investigator — University of Michigan
Locations (1):
- Chronic Pain and Fatigue Research Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aday JS, McAfee J, Conroy DA, Hosanagar A, Tarnal V, Weston C, Scott K, Horowitz D, Geller J, Harte SE, Pouyan N, Glynos NG, Baker AK, Guss J, Davis AK, Burgess HJ, Mashour GA, Clauw DJ, Boehnke KF. Preliminary safety and effectiveness of psilocybin-assisted therapy in adults with fibromyalgia: an open-label pilot clinical trial. Front Pain Res (Lausanne). 2025 Mar 18;6:1527783. doi: 10.3389/fpain.2025.1527783. eCollection 2025. PMID 40171515

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 17 participants were consented for this trial, 10 of whom were screen fails. Of the 7 remaining participants, 5 received the intervention and completed the trial.
Groups:
- Open Label Dosing Arm (15mg and 25mg): This is an open-label study, and participants who meet the inclusion and exclusion criteria will be eligible and invited to enroll. Enrolled participants are planned to receive 2 doses of psilocybin: a 15 mg dose followed 2 weeks later by a 25 mg dose. The total planned duration of the study for an individual participant from screening to last follow-up is approximately 8 months.
  Psilocybin: Two oral doses of psilocybin in a capsule formulation taken approximately 2 weeks apart.
  Psychotherapy: 1. Pre-dose preparatory sessions; 2. Dosing day monitoring; and, 3. Post-dose integration sessions.
Period: Overall Study
Arm/Group | Open Label Dosing Arm (15mg and 25mg)
Started | 7
Received 15 mg Dose (Day 22) | 5
Received Second 15 mg Dose (Day 36) | 1
Received 25 mg Dose (Day 36) | 4
Completed | 5
Not Completed | 2
Not completed — Concerns about participant ability to follow study procedures | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: 17 participants were recruited for the trial, 10 of whom were screen fails. Of the 7 remaining participants, 5 received the intervention and completed the trial.
Arm/Group | Open Label Dosing Arm (15mg and 25mg)
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.06 (14.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Heart Rate Beats Per Minute (BPM) - First Dose (15 mg)
Description: BPM was measured before TRP-8802 capsule administration and at 30, 60, 90, 120, 180, 240, 300, and 360 minutes after capsule administration.
Time Frame: Day 22 Pre-Dose (Baseline) and at 30, 60, 90, 120, 180, 240, 300, and 360 minutes post-dose
Population: Results reflect the participants who completed the trial.
Measure: Median (Full Range); unit: Heart beats per minute
Arm/Group | Open Label Dosing Arm (15mg and 25mg)
Number analyzed (Participants) | 5
Heart beats per minute
  Baseline (before capsule administration) | 76 [64 to 85]
  30 minutes after capsule administration | 67 [59 to 81]
  60 minutes after capsule administration | 67 [61 to 83]
  90 minutes after capsule administration | 68 [61 to 88]
  120 minutes after capsule administration | 74 [65 to 87]
  180 minutes after capsule administration | 83 [63 to 87]
  240 minutes after capsule administration | 79 [67 to 94]
  300 minutes after capsule administration | 82 [75 to 88]
  360 minutes after capsule administration | 72 [71 to 87]

2. Primary Outcome: Heart Rate Beats Per Minute (BPM) - Second Dose (25 mg)
Description: as for outcome 1
Time Frame: Day 36 Pre-Dose (Baseline) and at 30, 60, 90, 120, 180, 240, 300, and 360 minutes post-dose
Population: Results reflect the participants who completed the trial. 1 participant elected to take a second 15 mg dose rather than the 25 mg dose. That participant's data was included in the results for this outcome.
Measure: Median (Full Range); unit: Heart beats per minute
Arm/Group | Open Label Dosing Arm (15mg and 25mg)
Number analyzed (Participants) | 5
Heart beats per minute
  Baseline (before capsule administration) | 75 [70 to 95]
  30 minutes after capsule administration | 85 [57 to 88]
  60 minutes after capsule administration | 82 [57 to 90]
  90 minutes after capsule administration | 80 [56 to 86]
  120 minutes after capsule administration | 80 [56 to 88]
  180 minutes after capsule administration | 75 [60 to 101]
  240 minutes after capsule administration | 80 [62 to 106]
  300 minutes after capsule administration | 86 [64 to 115]
  360 minutes after capsule administration | 76 [61 to 106]

3. Primary Outcome: Blood Pressure (BP) - First Dose (15 mg) - Systolic
Description: Systolic BP was measured in millimeters of mercury (mm Hg) before TRP-8802 capsule administration and at 30, 60, 90, 120, 180, 240, 300, and 360 minutes after capsule administration. Systolic BP greater than 200 for more than 15 minutes was considered to be an adverse event.
Time Frame: Day 22 Pre-Dose (Baseline) and at 30, 60, 90, 120, 180, 240, 300, and 360 minutes post-dose
Population: Results reflect the participants who completed the trial.
Measure: Median (Full Range); unit: mm Hg
Arm/Group | Open Label Dosing Arm (15mg and 25mg)
Number analyzed (Participants) | 5
mm Hg
  Baseline (before capsule administration) | 133 [122 to 141]
  30 minutes after capsule administration | 126 [110 to 139]
  60 minutes after capsule administration | 131 [124 to 159]
  90 minutes after capsule administration | 137 [124 to 145]
  120 minutes after capsule administration | 131 [121 to 181]
  180 minutes after capsule administration | 141 [120 to 147]
  240 minutes after capsule administration | 130 [119 to 143]
  300 minutes after capsule administration | 128 [113 to 166]
  360 minutes after capsule administration | 135 [125 to 154]

4. Primary Outcome: Blood Pressure (BP) - Second Dose (25 mg) - Systolic
Description: BP was measured in millimeters of mercury (mm Hg) before TRP-8802 capsule administration and at 30, 60, 90, 120, 180, 240, 300, and 360 minutes after capsule administration. Systolic BP greater than 200 for more than 15 minutes was considered to be an adverse event.
Time Frame: Day 36 Pre-Dose (Baseline) and at 30, 60, 90, 120, 180, 240, 300, and 360 minutes post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: mm Hg
Arm/Group | Open Label Dosing Arm (15mg and 25mg)
Number analyzed (Participants) | 5
mm Hg
  Baseline (before capsule administration) | 135 [114 to 147]
  30 minutes after capsule administration | 123 [112 to 167]
  60 minutes after capsule administration | 140 [117 to 183]
  90 minutes after capsule administration | 141 [106 to 180]
  120 minutes after capsule administration | 127 [114 to 171]
  180 minutes after capsule administration | 142 [126 to 178]
  240 minutes after capsule administration | 134 [116 to 151]
  300 minutes after capsule administration | 134 [128 to 141]
  360 minutes after capsule administration | 141 [108 to 151]

5. Primary Outcome: Blood Pressure (BP) - First Dose (15 mg) - Diastolic
Description: Diastolic BP was measured in millimeters of mercury (mm Hg) before TRP-8802 capsule administration and at 30, 60, 90, 120, 180, 240, 300, and 360 minutes after capsule administration. BP greater than 110 diastolic for more than 15 minutes was considered to be an adverse event.
Time Frame: Day 22 Pre-Dose (Baseline) and at 30, 60, 90, 120, 180, 240, 300, and 360 minutes post-dose
Population: Results reflect the participants who completed the trial.
Measure: Median (Full Range); unit: mm Hg
Arm/Group | Open Label Dosing Arm (15mg and 25mg)
Number analyzed (Participants) | 5
mm Hg
  Baseline (before capsule administration) | 81 [64 to 85]
  30 minutes after capsule administration | 76 [68 to 78]
  60 minutes after capsule administration | 74 [64 to 79]
  90 minutes after capsule administration | 75 [68 to 87]
  120 minutes after capsule administration | 75 [67 to 86]
  180 minutes after capsule administration | 78 [67 to 80]
  240 minutes after capsule administration | 64 [62 to 81]
  300 minutes after capsule administration | 67 [61 to 80]
  360 minutes after capsule administration | 84 [72 to 86]

6. Primary Outcome: Blood Pressure (BP) - Second Dose (25 mg) - Diastolic
Description: as for outcome 5
Time Frame: Day 36 Pre-Dose (Baseline) and at 30, 60, 90, 120, 180, 240, 300, and 360 minutes post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: mm Hg
Arm/Group | Open Label Dosing Arm (15mg and 25mg)
Number analyzed (Participants) | 5
mm Hg
  Baseline (before capsule administration) | 82 [70 to 95]
  30 minutes after capsule administration | 65 [64 to 79]
  60 minutes after capsule administration | 74 [61 to 87]
  90 minutes after capsule administration | 74 [59 to 82]
  120 minutes after capsule administration | 70 [56 to 83]
  180 minutes after capsule administration | 78 [64 to 83]
  240 minutes after capsule administration | 80 [70 to 81]
  300 minutes after capsule administration | 69 [63 to 88]
  360 minutes after capsule administration | 80 [55 to 92]

7. Primary Outcome: Adverse Events (AE) Incidence
Description: Results reflect the total number of all adverse events that occurred during the trial.
Time Frame: Day 1 through Day 64
Population: Results reflect the participants who completed the trial.
Measure: Number; unit: Adverse Events
Arm/Group | Open Label Dosing Arm (15mg and 25mg)
Number analyzed (Participants) | 5
Adverse Events | 20

8. Secondary Outcome: Change in Pain Interference
Description: Pain interference is the degree to which pain affects important aspects of an individual's life, such as social, cognitive, and physical activities. Pain interference was assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) pain interference scale from the PROMIS-29+2 Profile v2.1 (PROPr). The raw scores were converted to standardized T-scores, with 50 as the population mean with a standard deviation of 10, and higher scores indicating worse pain interference.
Time Frame: Day 1 and Day 64
Population: Results reflect the participants who completed the trial.
Measure: Mean (Full Range); unit: t-score
Arm/Group | Open Label Dosing Arm (15mg and 25mg)
Number analyzed (Participants) | 5
t-score
  Pre capsule administration (Day 1) | 62.5 [57.1 to 66.6]
  Post capsule administration (Day 64) | 53.1 [41.6 to 57.1]

9. Secondary Outcome: Sleep Disturbance
Description: Sleep disturbance included assessment of sleep quality, perceived ability to fall and stay asleep, satisfaction of sleep, and depth of sleep. Sleep disturbance was measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance Short Form 8b. The raw scores were converted to standardized T-scores, with 50 as the population mean with a standard deviation of 10, and higher scores indicating worse sleep disturbance.
Time Frame: Day 1 and Day 64
Population: Results reflect the participants who completed the trial.
Measure: Mean (Full Range); unit: t-score
Arm/Group | Open Label Dosing Arm (15mg and 25mg)
Number analyzed (Participants) | 5
t-score
  Pre capsule administration (Day 1) | 58.2 [50.1 to 62.6]
  Post capsule administration (Day 64) | 51.1 [47.9 to 55.3]

10. Secondary Outcome: Chronic Pain Acceptance
Description: Chronic Pain Acceptance was measured using that Chronic Pain Acceptance Questionnaire-8 (CPAQ-8) that assessed activity engagement and pain willingness (e.g., recognizing that trying to avoid or control pain may be maladaptive for chronic pain). The lowest possible score was 0 (full chronic pain acceptance) and the highest possible score was 48 (no chronic pain acceptance).
Time Frame: Day 1 and Day 64
Population: Results reflect the participants who completed the trial.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Open Label Dosing Arm (15mg and 25mg)
Number analyzed (Participants) | 5
score on a scale
  Pre capsule administration (Day 1) | 28.4 [23 to 31]
  Post capsule administration (Day 64) | 30.4 [26 to 35]

11. Secondary Outcome: Patient Global Impression of Change (PGI-C)
Description: The PGI-C was a questionnaire that gauged the participant's response to medical interventions using a 7-point Likert scale ranging from 1 to 7 with 1 being "very much improved" and 7 being "very much worse".
Time Frame: Day 64
Population: Results reflect the participants who completed the trial.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Open Label Dosing Arm (15mg and 25mg)
Number analyzed (Participants) | 5
Score on a scale | 2 [1 to 3]

12. Secondary Outcome: Chronic Pain Intensity Between Groups in the Study Period
Description: Aggregated worst pain intensity scale from 0 (no pain) to 10 (highest pain possible) during 7-day epochs from day 1 through day 64. Participants' scores from Days 1-7 and Days 57-63 were compared.
Time Frame: Days 1-7 & Days 57-63
Population: Results reflect the participants who completed the trial.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Open Label Dosing Arm (15mg and 25mg)
Number analyzed (Participants) | 5
score on a scale
  Days 1-7 | 4.9 [3.7 to 5.9]
  Days 57-63 | 2.5 [1.1 to 2.7]

ADVERSE EVENTS:
Time Frame: Up to 8 months
Description: Results reflect the participants who received the intervention and completed the trial. As shown in the milestones under the Participant Flow, 1 participant did not receive the 25 mg dose and opted to receive a second 15 mg dose. Therefore, that participant is not included in the denominators for AEs involving the 25 mg dose.
Groups:
- Open Label Dosing Arm (15mg and 25mg): Enrolled participants received 2 doses of psilocybin: a 15 mg dose followed 2 weeks later by a second dose, which was planned to be 25 mg. 1 participant elected the second dose to be 15 mg instead. The total planned duration of the study for an individual participant from screening through pre-dose preparatory sessions to last follow-up was approximately 8 months.
  Psilocybin: Two oral doses of psilocybin in a capsule formulation taken approximately 2 weeks apart.
  Psychotherapy: 1. Pre-dose preparatory sessions; 2. Dosing day monitoring; and 3. Post-dose integration sessions.
Arm/Group | Open Label Dosing Arm (15mg and 25mg)
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 4/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Open Label Dosing Arm (15mg and 25mg) (N=5)
Fatigue (Pre-Dose) (Endocrine disorders) | 1
Diarrhea (following 15 mg dose) (Gastrointestinal disorders) | 2
Diarrhea (following 25 mg dose) (Gastrointestinal disorders) | 1/4
Stomach Ache (following 15 mg dose) (Gastrointestinal disorders) | 1
Vomiting (following 25 mg dose) (Gastrointestinal disorders) | 1/4 — 1 participant did not receive the 25 mg dose
Sore Throat (following 25 mg dose) (General disorders) | 1/4 — 1 participant did not receive the 25 mg dose
Back Ache (Pre-Dose) (Musculoskeletal and connective tissue disorders) | 1
Back Ache (following 15 mg dose) (Musculoskeletal and connective tissue disorders) | 1
Body Aches (following 25 mg dose) (Musculoskeletal and connective tissue disorders) | 1/4 — 1 participant did not receive the 25 mg dose
Jaw Pain (temporomandibular joint dysfunction [TMJ]) (Pre-dose) (Musculoskeletal and connective tissue disorders) | 1
Leg Throbbing (following 15 mg dose) (Musculoskeletal and connective tissue disorders) | 1 — 1 participant did not receive the 25 mg dose
Tight Left Side of Neck (Pre-Dose) (Musculoskeletal and connective tissue disorders) | 1
Tight Left Side of Neck (following 25 mg dose) (Musculoskeletal and connective tissue disorders) | 1/4 — 1 participant did not receive the 25 mg dose
Chills (following 25 mg dose) (Nervous system disorders) | 1/4 — 1 participant did not receive the 25 mg dose
Fever (following 25 mg dose) (Nervous system disorders) | 1/4 — 1 participant did not receive the 25 mg dose
Headache (Following 15 mg dose) (Nervous system disorders) | 3
Headache (Pre-Dose) (Nervous system disorders) | 1
Headache (following 25 mg dose) (Nervous system disorders) | 3/4 — 1 participant did not receive the 25 mg dose
Migraine (following 15 mg dose) (Nervous system disorders) | 1
Sinus Pressure (following 25 mg dose) (Respiratory, thoracic and mediastinal disorders) | 1/4 — 1 participant did not receive the 25 mg dose

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-28): https://cdn.clinicaltrials.gov/large-docs/62/NCT05128162/Prot_SAP_001.pdf